CLINICAL TRIAL: NCT07296094
Title: Psilocybin-Assisted Psychotherapy for the Treatment of Severe Alcohol Use Disorder: A Double-Blind, Dose-Comparison Concurrent Control Randomized Trial
Brief Title: Psilocybin-Assisted Psychotherapy for the Treatment of Severe Alcohol Use Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joji Suzuki, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P002909
Record Dates: First submitted 2025-12-12; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol use disorder; psilocybin; inpatient withdrawal management; psychedelic
MeSH Terms: conditions — Alcoholism | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: This study uses a double-blind, parallel-group, dose-comparison concurrent control, randomized trial design. Participants are randomly assigned in a 1:1 ratio to receive two sessions of either a full dose (30 mg with optional escalation to 40 mg) or a low dose (10 mg with optional escalation to 15 mg). All participants receive two dosing sessions four weeks apart, along with a standardized psychotherapy protocol delivered before, during, and after each session. Outcomes are assessed repeatedly from baseline through 48 weeks after the second dose, allowing evaluation of both clinical effects and mechanistic changes over time.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial uses double-blind masking. Participants, therapists, clinical staff present during dosing sessions, outcome assessors, and study investigators are all masked to treatment assignment. The psilocybin doses are prepared and dispensed by unmasked pharmacy personnel who have no contact with participants and no role in assessments or data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dose Psilocybin (Active Comparator): Participants randomized to this arm receive psilocybin in capsule form at a dose of 10 mg during the first dosing session, with the option to increase to 15 mg at the second session. Doses are administered orally under direct supervision in a controlled clinical setting and paired with the same standardized psychotherapy protocol used in the high-dose arm. Participants complete two dosing sessions four weeks apart and receive ongoing support from a peer recovery coach and optional outpatient addiction treatment.
  Interventions: Drug: Psilocybin
- Full Dose Psilocybin (Experimental): Participants randomized to this arm receive psilocybin in capsule form at a dose of 30 mg during the first dosing session, with the option to increase to 40 mg at the second session. Doses are administered orally under direct supervision in a controlled clinical setting and paired with a standardized psychotherapy protocol, including preparatory and integration sessions. All participants complete two dosing sessions spaced four weeks apart and receive ongoing support from a peer recovery coach and optional outpatient addiction treatment.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin is administered in oral capsule form during two dosing sessions held four weeks apart. Each session occurs in a controlled clinical environment with continuous monitoring by trained study therapists. Participants receive a standardized psychotherapy protocol that includes preparatory sessions before dosing and integration sessions afterward. The randomized dosing schedule includes either 10 mg with optional escalation to 15 mg or 30 mg with optional escalation to 40 mg for the second session. All participants also receive support from a peer recovery coach and are offered ongoing outpatient addiction treatment throughout the study period.

SUMMARY:
This study aims to determine the safety and preliminary efficacy of psilocybin-assisted psychotherapy in improving alcohol-related outcomes among adults with severe alcohol use disorder in a a double-blind, dose-comparison concurrent control, randomized trial. Participants will undergo structured psychotherapy and will be randomized to two psilocybin sessions to receive either a full dose (30mg or 40mg) or low dose (10mg or 15mg).

DETAILED DESCRIPTION:
This study is a double-blind, dose-comparison concurrent control randomized trial designed to evaluate the effects of psilocybin-assisted psychotherapy on alcohol-related outcomes, neurocognitive processes related to craving and stress, and neural circuits involved in reward and regulation among adults with severe alcohol use disorder (AUD). Participants are recruited up to 3 months after completing inpatient alcohol withdrawal treatment to ensure medical stabilization prior to psilocybin administration. The study examines both preliminary efficacy and safety while also exploring mechanistic pathways through behavioral assessments and functional neuroimaging.

Participants (N=36) are randomized in a 1:1 ratio to receive either a full-dose psilocybin (30 mg, with option to escalate to 40 mg on the second session) or a low-dose (10 mg, with option to escalate to 15 mg on the second session). All participants complete two dosing sessions spaced four weeks apart. The psychotherapy is delivered by a dyad of trained therapists before, during, and after the dosing sessions and is based on established therapeutic frameworks used in prior psilocybin-assisted therapy trials. The aim of the therapeutic support is to prepare participants for the psilocybin experience, facilitate psychological processing during and after dosing, and support integration of insights into daily life.A peer recovery coach is integrated into the study to support relapse prevention, enhance coping skills, and encourage engagement in ongoing addiction treatment. All participants are offered follow-up services at the institution's outpatient addiction treatment program (including the BWH Bridge Clinic), regardless of study arm. This combination of medical oversight, psychotherapy, and recovery support reflects an effort to embed the intervention within real-world addiction care settings.

Alcohol-related outcomes are assessed repeatedly from baseline through 48 weeks after the second dosing session. The primary clinical outcome is the percentage of heavy drinking days during the 24-week follow-up period, measured using Timeline Follow-Back. Secondary alcohol outcomes include drinking quantity and frequency, relapse timing, direct alcohol biomarkers (phosphatidylethanol and ethylglucuronide), withdrawal symptoms, treatment expectancy, blinding integrity, and quality of life measures. Additional exploratory outcomes assess peer support engagement and 12-step attendance.

Safety is evaluated throughout the study using structured assessments of adverse events, vital signs, and mood and anxiety symptoms. Because participants have severe AUD and recent withdrawal treatment, careful medical screening is conducted prior to each dosing session. The study includes multiple follow-up assessments up to 48 weeks after the second psilocybin dose, allowing characterization of both acute and longer-term safety.

Two mechanistic components are incorporated. First, neurocognitive tasks assess cue-induced craving, attentional bias, stress reactivity, delayed discount, decision making, and distress tolerance. These measures evaluate whether psilocybin influences cognitive and affective processes known to contribute to alcohol use and relapse. Second, participants complete two fMRI scans-first within one week prior to the first dosing session and the second within one week after the second dosing session. The fMRI tasks evaluate neural response to alcohol-related cues and the ability to down-regulate craving, focusing on the nucleus accumbens (NAcc) and dorsolateral prefrontal cortex (DLPFC). Connectivity analyses examine changes in functional coupling between these regions during alcohol cue processing.

Together, these approaches allow the study to evaluate whether full-dose psilocybin, compared to low-dose, produces greater reductions in heavy drinking and craving, whether the treatment is safe and tolerable for individuals with severe AUD, and whether changes in cognitive, emotional, and neural functioning help explain clinical outcomes. By recruiting individuals immediately following inpatient detoxification, the study also examines the feasibility of incorporating psilocybin-assisted therapy into a critical window of early recovery. Results will inform whether a larger, fully powered clinical trial is justified and will contribute to the broader understanding of psilocybin's therapeutic potential in alcohol use disorder.

ELIGIBILITY:
To be eligible, individuals must be:

* English speaking adults between ages 18 and 65
* Diagnosis of DSM5 AUD, severe
* Completion of inpatient withdrawal management (i.e. "detox") for AUD within 90 days of enrollment
* Amenable to attending all psychotherapy and study visits at BWH CCI
* Able to identify an individual who can act as points of contact during the trial
* Have a friend or family member who can bring the participant home after the psilocybin sessions and stay overnight

Individuals with any of the following will be excluded:

* Any personal history of a psychotic disorder (schizophrenia, schizoaffective disorder, brief psychotic disorder, delusional disorder, schizophreniform disorder, substance-induced psychotic disorder or major depression with psychotic features) or any bipolar-spectrum disorder
* Participants with a family history of first-degree relatives with psychotic disorder or bipolar-spectrum disorder
* Participants who have a significant suicide risk as defined by current suicidal ideation (Columbia-Suicide Severity Rating Scale (C-SSRS) score 2 to 5) and/or recent (within the past 6 months) active suicidal ideation (C-SSRS score 4 or 5)
* Participants who have a history of significant or serious adverse reaction to classic psychedelics
* Homicidality within the last six months
* History of DSM5 hallucinogen use disorder
* Positive blood alcohol level at screening
* Need for inpatient withdrawal management for alcohol at the time of screening
* Current DSM5 opioid, cocaine, stimulant or sedative/hypnotic use disorder
* Systolic blood pressure persistently above 165mmHg during screening
* History of hypersensitivity to psilocybin
* Use of psilocybin or other psychedelics with 5-HT2B activity in the prior 12 months
* Significant EKG abnormalities including QTc prolongation defined as >450 ms for men and women, or a diagnosis or family history of Long QT syndrome.
* History of any cardiac valvulopathy that raises the risk for participation as determined by the cardiology consultant
* History of intracranial mass or bleed, seizure disorder other than alcohol withdrawal seizures, liver cirrhosis, renal failure, obstructive lung disease requiring supplemental oxygen, hyperthyroidism, narrow-angle glaucoma, uncontrolled cardiac arrythmias, heart failure
* History of head trauma, stroke, or myocardial infarction in one year prior to enrollment.
* Expected to require surgical treatment at any point during the trial
* Liver dysfunction with LFTs > 3x upper normal limit at screening and Total bilirubin > 2.5x the upper normal limit
* MRI contraindications (other ferromagnetic implants, body weight greater than 550 lbs., etc.)
* Pregnant or breastfeeding
* High risk for adverse emotional or behavioral reaction based on the opinion of the study investigators such as evidence of a personality disorder
* Currently taking medications with serotonergic activity (other than SSRIs/SNRIs); inhibitors of UGT1A9, UGT1A10, MAO, and aldehyde or alcohol dehydrogenase; antipsychotics (e.g., first and second generation); mood stabilizers (e.g., lithium, valproic acid); or significant inhibitors of UGT enzymes that metabolize psilocin
* Selective serotonergic reuptake inhibitors and serotonin and norepinephrine reuptake inhibitors are allowed if participants have been on stable doses of the medication(s) for at least 30 days prior to enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Percent Heavy Drinking Days | Weeks 0-24 following the first psilocybin dosing session.
  Percent Heavy Drinking Days (PHDD) is defined as the percentage of days in which participants engage in heavy drinking, calculated using the Timeline Follow-Back (TLFB) method. Heavy drinking is defined using NIAAA criteria (≥4 drinks/day for women; ≥5 drinks/day for men). PHDD will be analyzed as a continuous outcome to compare change over time between the full-dose and low-dose psilocybin groups.
Adverse effects | 1, 2, 4, 8, 16, 24 and 48 weeks after receiving the second dose of the psilocybin treatment.
  We will utilize the Patient-Rated Inventory of Side Effects to assess the frequency and severity of adverse effects.
Cue-Induced Craving Response | Measured at baseline, 4 and 24 weeks after the second psilocybin treatment.
  Craving intensity elicited by alcohol-related visual cues during a standardized cue-reactivity task as measured using a visual analog scale. The scale is titled Cue induced Craving scale and is measured from 0-10, 0 being Not at all and 10 being extremely craving. A higher score indicates more craving of the substance shown.
Neural Response and Connectivity Changes measured by fMRI | 1 week before and 1 week after the second psilocybin session
  BOLD response in the nucleus accumbens (NAcc) to alcohol-related images during craving.
Neural Response and Connectivity Changes measured by fMRI | 1 week before and 1 week after the second psilocybin session
  BOLD response in the dorsolateral prefrontal cortex (DLPFC) during down-regulation of craving.
Neural Response and Connectivity Changes measured by fMRI | 1 week before and 1 week after the second psilocybin session
  NAcc-DLPFC functional connectivity during alcohol cue processing.

SECONDARY OUTCOMES:
Percent Days Abstinent | Baseline to Weeks 24
  Percentage of days with no alcohol use, based on TLFB.
Drinks Per Drinking Day | Baseline to Week 24
  Number of standard drinks consumed on days with any drinking, assessed using the Timeline Follow-Back (TLFB) method.
Vital signs | Baseline to Week 48
  Blood pressure
MEQ30 - Mystical Experience Questionnaire. | Visit 6 & 10 (about 4 weeks in between visits 6 and 10)
  The Mystical Experience Questionnaire (MEQ-30) is a 30-item self-report measure assessing the intensity of mystical-type experiences during a psychedelic session. Scores are calculated for Transcendence, Positive Mood, Ineffability, Mystical experience, and as a total score, with each expressed as a percentage of the maximum possible score. Higher percentages indicate more intense and complete mystical experiences.
Altered states of consciousness | Immediately after each drug session
  5-dimensional Altered States of Consciousness questionnaire
Distress Tolerance | Measured at baseline, 4 and 24 weeks after the second psilocybin treatment.
  Mirror Tracing Persistence Task- Assesses distress tolerance.
Days to Relapse | Baseline to Week 48
  Number of days from first psilocybin dose to first consumption of alcohol following inpatient withdrawal treatment.
Days to First Heavy Drinking Day | Baseline to Week 48
  Number of days from first psilocybin dose to first heavy drinking episode, defined using NIAAA criteria.
WHO Drinking Risk Level | Baseline; Weeks 1, 2, 4, 8, 16, 24, and 48
  Change in WHO alcohol risk classification categories based on self-reported alcohol consumption.
Phosphatidylethanol (PEth) Levels | Baseline; Weeks 4, 8, 24, and 48
  Blood biomarker of recent alcohol use measured via PEth concentration.
Ethylglucuronide (EtG) Levels | Baseline; Weeks 4, 8, 24, and 48
  Urine biomarker of recent alcohol consumption measured via EtG levels.
Alcohol Withdrawal Severity | Baseline to Week 24
  The Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar) is a clinician-administered scale used to assess the severity of alcohol withdrawal symptoms. It includes 10 items evaluating symptoms such as tremor, anxiety, agitation, nausea, and hallucinations, with total scores ranging from 0 to 67. Higher scores indicate more severe withdrawal and guide clinical management and treatment decisions.
Treatment Expectancy: Set and Setting (Stanford Expectancy Treatment Scale; SETS) | Visit 1- Baseline visit
  Participant expectations regarding treatment benefit measured prior to any psilocybin dosing. The Stanford Expectancy Treatment Scale (SETS) is a self-report measure assessing participants' expectations, mindset ("set"), and perceptions of the treatment context ("setting") prior to an intervention. It evaluates beliefs about treatment credibility, anticipated benefits, and the therapeutic environment. Higher scores indicate more positive expectations and a more supportive perceived setting.
Assessment of Blinding | Visit 6 and 10, 4 weeks between
  Participant and clinician guesses regarding dose assignment to evaluate masking integrity.
Alcohol Craving (Penn Alcohol Craving Scale; PACS | Baseline; Weeks 1, 2, 4, 8, 16, 24, and 48
  he Penn Alcohol Craving Scale (PACS) is a 5-item self-report measure assessing the frequency, intensity, and duration of alcohol craving over the past week. Total scores range from 0 to 30. Higher scores indicate greater alcohol craving severity.
Quality of Life (WHOQOL-BREF) | Baseline; Weeks 8, 24, and 48
  The World Health Organization Quality of Life-BREF (WHOQOL-BREF) is a self-report measure assessing overall quality of life across physical health, psychological health, social relationships, and environment. Scores are calculated for each domain and transformed to standardized scales. Higher scores indicate better perceived quality of life.
Peer Support Engagement | Baseline to Week 48
  Frequency and extent of interactions with the peer recovery coach across the study period.
12-Step Meeting Attendance | Baseline to Week 48
  Self-reported attendance at Alcoholics Anonymous or other mutual-help meetings.
Depression Severity (PHQ-9) | Baseline to Week 48
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report measure assessing depressive symptom severity over the past two weeks. Total scores range from 0 to 27. Higher scores indicate greater severity of depressive symptoms.
Anxiety Severity (GAD-7) | Baseline to Week 48
  The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item self-report measure assessing anxiety symptom severity over the past two weeks. Total scores range from 0 to 21. Higher scores indicate greater anxiety severity
Suicidality (C-SSRS) | Baseline to Week 48
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinician-administered measure assessing the severity and intensity of suicidal ideation and behavior. It evaluates the presence, frequency, and lethality of suicidal thoughts and actions over specified time frames. Higher severity ratings indicate greater suicide risk and inform clinical monitoring and intervention.
Liver Function Tests | Baseline; routine follow-up through Week 48
  Laboratory evaluation of hepatic safety using standard liver enzyme markers.
Hospital Readmission | Baseline to Week 48
  Documentation of any all-cause hospital readmissions during the follow-up period.
Attentional Bias to Alcohol Cues (Visual Probe Task) | Assessed using the Visual Probe Task (VPT), which measures attentional bias through reaction time differences when responding to probes replacing alcohol-related vs. neutral stimuli.
  Baseline; Weeks 4 and 24 after the second psilocybin session
Delayed Discounting (Monetary Choice Questionnaire) | Baseline; Weeks 4 and 24 after the second psilocybin session
  Measured using the Monetary Choice Questionnaire, which presents choices between smaller immediate rewards and larger delayed rewards. The calculated discount rate (k-value) reflects impulsive choice and reward valuation.
Decision-Making Performance (Iowa Gambling Task) | Baseline; Weeks 4 and 24 after the second psilocybin session
  Measured using the Iowa Gambling Task (IGT). Participants select cards from decks with varying reward and penalty structures. Performance reflects learning from feedback and risk-sensitive decision making.
Vital signs | Baseline to Week 48
  Heart rate will be measured.
Vital signs | Baseline to Week 48
  Temperature will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Joji Suzuki, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States